CLINICAL TRIAL: NCT04161612
Title: Sleep Quality in Patients With Spinal Cord Injury
Brief Title: Sleep Quality & Spinal Cord Injury
Acronym: SLP
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Tuğba Aydın, Researcher, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: IstPMRTRH-SLP
Record Dates: First submitted 2019-11-10; First posted 2019-11-13 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-11

CONDITIONS: Sleep Disorder
Keywords: Sleep quality
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders | interventions — Causality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Demographic characteristics, duration of spinal cord injury, spinal cord injurylevel, etiology, number of intermittent bladder catheterization (IC), number of night time — Observational clinical study
  Other Names: Modified Ashworth Scale, Beck Depression Index,Pittsburgh Sleep Quality Index, Epworth sleepiness scale, Barthel Index ,Douleur Neuropathique 4 questionnaire

SUMMARY:
The aim of the study was to evaluate sleep quality in patients with spinal cord injury; to investigate the relationship between sleep and spinal cord level, ambulation status, spasticity, quality of life, daily living activities, depressive status, neuropathic pain

DETAILED DESCRIPTION:
Since survival increases in patients with spinal cord injury, sleep disturbances, which are more frequently observed than the general population and have significant impacts on mortality, impair long-term quality of life.The aim of the study was to evaluate sleep quality in patients with spinal cord injury; to investigate the relationship between sleep and spinal cord level, ambulation status, spasticity, quality of life, daily living activities, depressive status, neuropathic pain Eighty patients with inpatient rehabilitation of spinal cord injury were included in the study.

Demographic characteristics, duration of spinal cord injury, spinal cord injury level, etiology, number of intermittent bladder catheterization (IC), number of night time IC, what time they slept, whether they woke up at night, classification of spinal cord injury were recorded.

Ambulation level with Functional Ambulation Classification (FAC), spasticity with Modified Ashworth Scale (MAS), depressive symptoms with Beck Depression Index (BDI), quality of life with short-form health survey (SF-36), sleep quality The Pittsburgh Sleep Quality Index (PSQI), daytime sleepiness Epworth sleepiness scale (ESS), activity of daily living with Barthel Index (BI), neuropathic pain were evaluated with the Douleur Neuropathique 4 questionnaire (DN4) scale.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age

Exclusion Criteria:

* Noncooperativity
* Traumatic brain injury or other cerebellar-related neurological disease such as hemiplegia.
* Patients with spinal shock

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with spinal cord injury hospitalized in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Functional Ambulation Classification (FAC) | 3 month
  FAC is defined in five stages according to the basic motor skills required for functional ambulation. FAC stage 0 is used to indicate non-functional ambulation, and stage 5 is used to indicate independent walking at each speed and on ground
Beck Depression Index (BI) | 3 month
  The severity of depressive symptoms was assessed using the BDI. This scale consists of 21 categories that evaluate the physical, emotional, cognitive, and motivational symptoms of depression, such as hopelessness, irritability, guilt, feelings of being punished, fatigue, and weight loss
Pittsburgh Sleep Quality Index (PSQI) | 3 month
  A questionnaire that assesses sleep quality and discomfort over the last 1 month. The total score is between 0-21. A higher total score indicates poor sleep quality. A score of 5 or more indicates poor sleep quality
Epworth sleepiness scale (ESS) | 3 month
  It is a simple questionnaire that measures daytime sleepiness level. Sleepiness is questioned in cases encountered in daily life. The total score is between 0-24. Daytime sleepiness increases as the score increases

SECONDARY OUTCOMES:
short-form health survey (SF-36) | 3 month
  SF-36 is a widely-used and well-documented health-related quality of life index. The SF-36 survey has eight sub-dimensions, including physical functioning, role limitations due to physical problems, pain, general health perception, mental health, role limitations due to emotional problems, vitality, and social functioning, which are evaluated individually
Douleur Neuropathique 4 questionnaire | 3 month
  Evaluate neuropathic pain. It consists of 10 questions. The maximum score is 10. Patients with a score of 4 or more are considered to have neuropathic pain

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA AYDIN, MD, Study Chair — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hulten VDT, Biering-Sorensen F, Jorgensen NR, Jennum PJ. A review of sleep research in patients with spinal cord injury. J Spinal Cord Med. 2020 Nov;43(6):775-796. doi: 10.1080/10790268.2018.1543925. Epub 2018 Dec 4. PMID 30513274
- [Background] Giannoccaro MP, Moghadam KK, Pizza F, Boriani S, Maraldi NM, Avoni P, Morreale A, Liguori R, Plazzi G. Sleep disorders in patients with spinal cord injury. Sleep Med Rev. 2013 Dec;17(6):399-409. doi: 10.1016/j.smrv.2012.12.005. Epub 2013 Apr 22. PMID 23618534